CLINICAL TRIAL: NCT01473342
Title: Mila Blooms Intervention Study: An App for Promoting Physical Activity and Health Diet Among Adolescent Survivors of Childhood Cancer
Brief Title: Mila Blooms Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00029579; 1R21CA155965-01A1 (NIH)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Childhood Cancer
Keywords: Healthy survivorship; Smartphones; Treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control & Intervention Phases (Other): The control phase will run for 8 weeks, including survey completion and accelerometer wear during Week 1 and Week 8. The intervention phase will run for the 9 weeks following the control phase; where participants are assigned a smartphone to interact with the Mila Blooms gaming app and integrated social network & receive weekly supportive coaching phone calls from study staff for 8 weeks (Week 9 - Week 16) followed by accelerometer wear & survey completion during the 9th and final week (Week 17).
  Interventions: Behavioral: Mila Blooms

INTERVENTIONS:
Behavioral: Mila Blooms — Behavioral intervention will be administered to 30 adolescent childhood cancer survivors & their parents (3 blocks of 10 survivor-parent(s) groups) who serve as their own controls. The intervention phase begins at Week 9 (immediately following the 8-week control phase) and runs for 9 weeks (Weeks 9 - 17). Adolescents are assigned a smartphone installed with the Mila Blooms app to use for the first 8 weeks (Weeks 9 - 16) of the intervention. The app integrates (1) tools for tracking health behaviors (e.g., diet, physical activity, etc.); (2) an avatar system to provide virtual rewards, and (3) a social network of users for support. As part of the intervention, adolescents will also receive weekly coaching phone calls from study staff to discuss areas of concern and to encourage goal-setting & participation. During the 9th week (Week 17), participants complete one final survey & accelerometer wear.

SUMMARY:
This study is focused on the development and pilot/feasibility testing of a smartphone application to promote a healthy diet, increase physical activity, and prevent weight gain in adolescent survivors of childhood cancer.

DETAILED DESCRIPTION:
While successful advancements in treatment for childhood Acute Lymphoblastic Leukemia (ALL) have resulted in a growing cohort of survivors, these survivors are at risk for a number of long-term health problems. This study proposes to develop and conduct feasibility testing for a smartphone application that would deliver a health behavior intervention to this population.

A formative phase focused on intervention and software development will be followed by a pilot/feasibility test of the intervention. Participants in the intervention will receive a customized study-designed mobile phone app with a social networking component in which users will be able to support one another. They will also receive personal support from a health counselor to help set goals and discuss areas of concern.

ELIGIBILITY:
Inclusion Criteria:

* Participants must speak & read/write fluent English;
* Adolescent must be between 12 and 19 years of age;
* Adolescent must have a previous diagnosis of childhood Acute Lymphoblastic Leukemia;
* Adolescent must be "off-therapy" (i.e., not in active or maintenance phase of cancer therapy) for at least 2 years;
* Adolescent must be cleared by his/her physician to participate (defined by obtaining a score of 80 or greater on the Karnofsky Scale as determined by their physician);
* Participants must have a working phone number;
* Adolescents must live at home with parents in order to facilitate parent involvement via support materials.

Exclusion Criteria:

* Physician reports that the patient has deficits in neurocognitive functioning that would preclude him/her from participating in a cognitive-oriented intervention;

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Mila Blooms Intervention at changing health behaviors. | ~9 weeks (from pre-intervention baseline to post-intervention follow-up)
  Test the feasibility of the Mila Blooms intervention at changing diet, physical activity, body mass index (BMI), and social cognitive mediators of health behavior change.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard F. Fuemmeler, Ph.D., MPH, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Dept. of Community and Family Medicine, Durham, North Carolina, United States